CLINICAL TRIAL: NCT00159224
Title: Study ACA-ARGE-04-001 "A Pilot, Open-Label Study Assessing Safety, Tolerability, Efficacy of a Simplified Lopinavir/Ritonavir Induction/Maintenance Therapy in HIV-Infected Subjects on Their First Protease Inhibitor-Based Regimen".
Brief Title: Induction-maintenance of Lopinavir/r in HIV-infected Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Huésped (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Pedro Cahn, Scientic Director, The Huesped Foundation, Fundación Huésped
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACA-ARGE-04-001
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: HIV Infections
Keywords: HIV; Simplification; Monotherapy; Treatment Naive; HIV-1 infection
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lopinavir/ritonavir monotherapy (Experimental): Patients with undetectable viral load while on 1st line ARV therapy will be randomized to the expermental arm: Lopinavir/ritonavir monotherapy
  Interventions: Drug: Lopinavir/ritonavir simplification strategy
- Lopinavir/Ritonavir plus 2 NRTIs (Active Comparator): Patients randomized to this arm will continue with standard of care triple therapy, based on Lopinavir/Ritonavir plus 2 NRTIs
  Interventions: Drug: Lopinavir/ritonavir simplification strategy

INTERVENTIONS:
Drug: Lopinavir/ritonavir simplification strategy — Simplification
  Other Names: Kaletra monotherapy simplification strategy

SUMMARY:
This study will assess the safety, tolerability and antiviral activity of a simplified PI-based treatment regimen (Kaletra,ä) compared to conventional HAART regimens in patients infected with HIV-1 who are on their first boosted-PI antiretroviral treatment regimen.

The potency of the antiviral activity of Kaletra has been clearly demonstrated in a wide spectrum of patients in a number of different clinical trials.6-9 The durable viral suppression seen after 4 years of therapy10 proves that it can provide effective, long-term treatment for people with HIV-1.

Data from one of these trials (M97-720),6 an ongoing Phase II study of lopinavir/ritonavir in combination with NRTIs suggests there may be a role for monoclass therapy with Kaletra in the treatment of HIV-1-infection.

ELIGIBILITY:
Inclusion Criteria:

* Subject has confirmed his or her willingness to participate in this study after being informed of all aspects of the trial that are relevant to his or her decision to take part, by signing and dating the IRB / IEC approved informed consent form.
* Subject is HIV positive and on their first antiretroviral treatment regimen, based on any two NRTIs plus lopinavir/ritonavir or a ritonavir-boosted PI combination. Subject must have had no previous exposure to other regimens.
* Subject has a viral load <50 copies/ml at the time of baseline evaluation for at least 6 months.
* Subject has a CD4 cell count ³ 100 cells/mm3.
* Subject is aged >18 years.
* Vital signs, physical examination and laboratory results do not exhibit evidence of acute illness.
* Subject has not been treated for an active opportunistic infection within 30 days of screening.
* If female, subject has a negative pregnancy test and agrees to use, for the duration of the study, a barrier method of birth control that has a history of proven reliability as judged by the investigator.
* Subject does not require and agrees not to take, for the duration of the study, any medication that is contraindicated with any of the antiretroviral drugs in their treatment regimen. The subject agrees not to take any medication, including over-the-counter medicine, alcohol, or recreational drugs without the knowledge and permission of the principal investigator

Exclusion Criteria:

* Subject has current uncontrolled substance abuse or psychiatric illness that could preclude compliance with the protocol.
* Subject has a viral load of > 50 copies/ml
* Subject is HBsAg +
* Subject has active tuberculosis or an opportunistic infection.
* Subject has active malignancy (except Kaposi's Sarcoma).
* Subject has liver failure as evidenced by ALT / AST > 5 x Upper Limit of Normal (ULN).
* Female subject is pregnant or lactating.
* Subject has received an investigational drug within 30 days prior to the initiation of the study.
* Subject has modified his/her antiretroviral therapy during the 3 months prior to baseline or is intending to do so during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients remaining undetectable below 50 copies/mL at 48 weeks | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pedro E Cahn, MD, PhD, Study Chair — Fundacion Huesped, Buenos Aires, Argentina; Julio SG Montaner, MD, Principal Investigator — University of British Columbia; Isabel L Cassetti, MD, Principal Investigator — Helios Salud, Buenos Aires, Argentina; Juan Sierra Madero, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricio Salvador Zurbaran, Mexico
Locations (4):
- Argentina (2):
  - Helios Salud, Buenos Aires
  - Fundacion Huesped, Buenos Aires
- University of British Columbia, Vancouver, British Columbia, Canada
- Instituto Nacional de Ciencias Medicas y Nutrición "Salvador Zubirán, Mexico City, Mexico

REFERENCES:
- [Derived] Cahn P, Montaner J, Junod P, Patterson P, Krolewiecki A, Andrade-Villanueva J, Cassetti I, Sierra-Madero J, Casiro AD, Bortolozzi R, Lupo SH, Longo N, Rampakakis E, Ackad N, Sampalis JS. Pilot, randomized study assessing safety, tolerability and efficacy of simplified LPV/r maintenance therapy in HIV patients on the 1 PI-based regimen. PLoS One. 2011;6(8):e23726. doi: 10.1371/journal.pone.0023726. Epub 2011 Aug 19. PMID 21886816